19 Versus 22-Gauge Fine Needle Biopsy (FNB) Needles for Endoscopic Ultrasound Guided Liver Biopsy (EUS-LB): A Prospective Pilot Study

NCT: NCT02967991 Date: August, 2016

## **Statistical Analysis**

This is a pilot study with a goal to obtain estimates to design a larger study. The precision, as measured by the half-width of a 95% confidence interval (CI) was used to select the sample size. It was assumed tissue adequacy for the control group was 88%. With a sample size of 40 subjects, the study is able to estimate a 95% CI with a half-width of 10% (i.e., 78%-98%).

Descriptive statistics were summarized for all demographic data including age, gender, and reason for EUS-LB. Continuous variables are reported as median and inter-quartile range, and categorical variables are shown as frequency and percentage. The 95% CI was estimated for the primary outcome of tissue adequacy. Even though this is a pilot study, statistical inference was performed to compare the wet and dry heparin groups to the control group. This was accomplished using McNemar's Chi square test for binary variables and the Wilcoxon Signed Rank test for continuous variables. Data analysis was performed using SAS v9.4 (SAS Institute Inc. Cary, NC). A p<0.05 was considered statistically significant